CLINICAL TRIAL: NCT06467435
Title: Evaluation of K9 in Subjects With Thyroid Eye Disease (TED)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Peter Timoney (Other)
Collaborators: Inflammasome Therapeutics (Industry)
Responsible Party: Sponsor-Investigator, Peter Timoney, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 94519
Record Dates: First submitted 2024-06-14; First posted 2024-06-21 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Thyroid Eye Disease
Keywords: Kamuvudine-9; K9
MeSH Terms: conditions — Graves Ophthalmopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Patients with Thyroid Eye Disease (TED) (Experimental): Participants receive a regimen of 96 mg tablets of K9 twice a day for 24 weeks
  Interventions: Drug: Kamuvudine-9
- Healthy Volunteers (Experimental): Participants receive one dose of 96 mg tablets of K9 based on weight
  Interventions: Drug: Kamuvudine-9

INTERVENTIONS:
Drug: Kamuvudine-9 — 96 mg tablets taken twice a day for 24 weeks
  Other Names: K9
  Arms: Patients with Thyroid Eye Disease (TED)
Drug: Kamuvudine-9 — 96 mg tablets taken once
  Other Names: K9
  Arms: Healthy Volunteers

SUMMARY:
The study is comprised of two cohorts. Cohort 1 will examine pharmacokinetics of K9 in 3 healthy volunteers over 24 hours. This cohort has been completed. Cohort 2 will involve up to 10 patients with TED. Patients will receive oral K9 BID for up to 24 weeks and will be followed up to a total of 26 weeks with a primary endpoint of safety.

ELIGIBILITY:
Inclusion Criteria:

Cohort 1

* Subject is willing and able to receive treatment and complete corresponding assessments as required by the protocol

Cohort 2

* Diagnosed with Thyroid Eye Disease (TED).
* Symptomatic TED diagnosed no more than 9 months earlier.
* Clinical Activity Score ≥ 3 (on 7 point scale) for the worse eye.
* Subject is willing and able to receive treatment and complete corresponding assessments as required by the protocol.

Exclusion Criteria:

Cohort 1

* Body weight less than 55 kg.
* History of any clinically significant medical disorders the principal investigator considers exclusionary, including (but not limited to), neuromuscular, hematological disease, immune deficiency state, respiratory disease, hepatic or gastrointestinal disease, neurological or psychiatric disease, ophthalmological disorders, neoplastic disease, renal or urinary tract diseases, or dermatological disease.
* Females who are pregnant, nursing, planning a pregnancy or who are of childbearing potential not using a reliable method of contraception.
* History or current evidence of hypersensitivity to any components of the study medication, as assessed by the investigator.
* Participation in any systemic experimental treatment or any other systemic investigational new drug within 6 weeks or 5 half-lives of the active ingredient (whichever is longer) prior to the start of study treatment. Clinical trials solely involving observation, over-the-counter vitamins, supplements, or diets are not exclusionary

Cohort 2

* Body weight less than 55 kg.
* Females who are pregnant, nursing, planning a pregnancy or who are of childbearing potential not using a reliable method of contraception.
* History or current evidence of hypersensitivity to any components of the study medication, as assessed by the investigator.
* Participation in any investigational drug or ocular device study within 30 days prior to the Day 1 Study Visit.
* History or current evidence of a medical condition that may, in the opinion of the investigator, preclude the safe administration of study medication or affect the results of the study.
* Participation in any systemic experimental treatment or any other systemic investigational new drug within 5 half-lives of the active ingredient prior to the start of study treatment. Clinical trials solely involving observation, over-the-counter vitamins, supplements, or diets are not exclusionary.
* History of use of teprotumumab (Tepezza), radiotherapy, or orbital surgery.
* History (last 6 weeks) of use of systemic immunosuppressants (e.g. mycophenolate), intravenous immunoglobulin, or plasmapheresis.
* Clinical activity score < 3
* Uncontrolled diabetes or hypertension
* History of mental / psychiatric disorder
* Hepatic dysfunction (Albumin (Alb), Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT) and Alkaline phosphates levels must be within normal range for eligibility)
* Renal impairment (Urea, Creatinine, and Glomerular Filtration Rate levels must be within normal range)
* Any baseline condition that the principal investigator considers exclusionary.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2024-11-06 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | 26 weeks
  Frequency of participants experiencing ocular or systemic adverse events.
plasma concentrations of K9 | Pharmacokinetic samples collected pre-dose and at 0.5, 1, 2, 3, 4, 6, 8, and 24 hours after dosing
  plasma concentrations measured after a single oral dose in healthy adults. For each of these time points 5 ml of blood will be drawn.

SECONDARY OUTCOMES:
Change in Standardized Patient Evaluation of Eye Dryness (SPEED) symptoms | Screening (Baseline), and Weeks 4, 14, and 24
  The SPEED Questionnaire will be used to track progression of dry eye symptoms. The SPEED questionnaire has eight questions. The frequency and severity of symptoms are rated on a numeric scale. Scores range from 0 to 28 with higher scores equating to more symptoms.
Change in Diplopia | Screening (Baseline), Day 1 Visit, and weeks 4, 14, and 24
  Diplopia is assessed by the Bahn-Gorman Scale. The Bahn-Gorman scale is a subjective grading scheme that uses a scale of 0-3 to assess the severity of diplopia. A higher score equates to more severe diplopia.
Change in Study Visit in Clinical Activity Score (CAS), | Screening (Baseline), Day 1 Visit, and weeks 4, 14, and 24
  Clinical Activity Score (7 point scale) with higher score equating to more symptoms
Change in proptosis | Screening (Baseline), Day 1 Visit, and weeks 4, 14, and 24
  Hertel exophthalmometry will be used to measure the globe position of the eye by calculating the distance from the lateral orbital rim to the surface of the cornea in millimeters (mm)
Change in Graves' ophthalmopathy-specific quality-of-life scale (GO-QOL) | Screening (Baseline) and weeks 4, 14, and 24
  The GO-QOL is a self-administered health-related QOL questionnaire specifically designed and validated in patients with TED. It includes 2 subscale GO-QOL scores: (1) visual functioning and (2) appearance-related, with the 2 weighted equally to create an overall score. Both the subscales and overall score are transformed to a scale of 0 to 100, 0 indicating worst health and 100 indicating best health.
Change in upper eyelid retraction | Screening (Baseline), Day 1 Visit, and weeks 4, 14, and 24
  upper eyelid retraction will be determined by measuring the margin reflex distance (MRD1) in millimeters. The MRD1 is the measurement in millimetres from the light reflex on the patient's cornea to the level of the centre of the upper eyelid margin, with the patient gazing in the primary position.
Change in lower eyelid retraction | Screening (Baseline), Day 1 Visit, and weeks 4, 14, and 24
  Lower eyelid retraction is measured by the distance from the inferior limbus to the lower eyelid, or by the margin reflex distance 2 (MRD2). The distance between the corneal light reflex to the central portion of the lower eyelid is measured in millimeters
Change in cell-based functional assays | Screening (Baseline), Day 1 Visit, and weeks 4,14, and 24
  measured by ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Peter Timoney, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No